CLINICAL TRIAL: NCT01693744
Title: The Relationship Between Pseudoexfoliation and Chronic Kidney Disease
Brief Title: Pseudoexfoliation and Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Corum State Hospital (Other)
Responsible Party: Principal Investigator, Leyla Niyaz, Ophthalmology Specialist, Corum State Hospital
Other Study IDs: LNiyaz
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Kidney Disease
Keywords: Pseudoexfoliation, chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dialysis patients: Patients with stage 5 chronic kidney disease undergoing haemodialysis
- Chronic kidney disease patients: Stage 1-4 Chronic kidney disease patients
- Control group: Patients with normal renal functions

SUMMARY:
Background: Pseudoexfoliation (PEX) is characterised by the deposition of fibrillar material in an eye structures and many other parts of the body including kidneys and blood vessels. As both PEX and chronic kidney disease (CKD) are associated with oxidative stress and endothelial dysfunction we studied if the risk of PEX was increased in patients with CKD.

Methods: Patients over age 40 with the diagnosis of CKD were included in the study. Chronic kidney disease was diagnosed as decreased glomerular filtration rate (GFR) of less than 60 mL/min/1.73 m². Study groups were arranged as group 1 consisting of HD receiving patients, group 2 consisting of stage 1-4 CKD patients and group 3 consisting of patients with normal kidney functions (control group). Demographic properties and the rate of PEX were evaluated and compaired between the groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic kidney disease stage 1-5

Exclusion Criteria:

* History of eye trauma or surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from nephrology clinic
Sampling Method: Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2011-10; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Prevalance of pseudoexfoliation in patients with chronic kidney disease | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Niyaz, M.D., Principal Investigator — Specialist in Ophthalmology
Locations (1):
- Corum State Hospital, Çorum, Turkey (Türkiye)